CLINICAL TRIAL: NCT01712425
Title: Safety and Immunogenicity of ChAdV63.HIVconsv and MVA.HIVconsv Candidate HIV-1 Vaccines in Recently HIV-1 Infected Individuals With Early Viral Suppression After Initiation of Antiretroviral Therapy (HAART)
Brief Title: Safety and Immunogenicity of ChAdV63.HIVconsv and MVA.HIVconsv Candidate HIV-1 Vaccines in Recently HIV-1 Infected Individuals
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: IrsiCaixa (Other)
Collaborators: Fundación FLS de Lucha Contra el Sida, las Enfermedades Infecciosas y la Promoción de la Salud y la Ciencia (Other); Hospital Clinic of Barcelona (Other); HIVACAT (Unknown); University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ChAd-MVA.HIVconsv-BCN01; 2011-000846-39 (EudraCT Number)
Record Dates: First submitted 2012-10-04; First posted 2012-10-23 (Estimated); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: HIV
Keywords: vaccine; recently HIV-1 infected individuals
MeSH Terms: interventions — PRIME protocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- 0-24 week prime/boost regimen (ARM A) (Experimental): Start antiretroviral treatment raltegravir + tenofovir/emtricitabine. ChAdV63.HIVcons and MVA.HIVconsv HIV-1 vaccines, delivered intramuscularly, 0-24 week prime/boost regimen
  Interventions: Biological: 0-24 week prime/boost regimen
- 0-8 week prime/boost regimen (ARM B) (Experimental): Start antiretroviral treatment raltegravir + tenofovir/emtricitabine. ChAdV63.HIVcons and MVA.HIVconsv HIV-1 vaccines, delivered intramuscularly, 0-8 week prime/boost regimen
  Interventions: Biological: 0-8 week prime/boost regimen
- Arm A control (ARM C) (No Intervention): Start antiretroviral treatment raltegravir + tenofovir/emtricitabine. Follow-up as in Arm A.
- Arm B control (ARM D) (No Intervention): Start antiretroviral treatment raltegravir + tenofovir/emtricitabine. Follow-up as in Arm B.

INTERVENTIONS:
Biological: 0-24 week prime/boost regimen — ChAdV63.HIVcons (5x10^10 vp) and MVA.HIVconsv (2x10^8 pfu) HIV-1 vaccines, delivered intramuscularly
  Other Names: ARM A
  Arms: 0-24 week prime/boost regimen (ARM A)
Biological: 0-8 week prime/boost regimen — ChAdV63.HIVcons (5x10^10 vp) and MVA.HIVconsv (2x10^8 pfu) HIV-1 vaccines, delivered intramuscularly
  Other Names: ARM B
  Arms: 0-8 week prime/boost regimen (ARM B)

SUMMARY:
The HIVconsv gene was constructed by assembling the 14 most conserved regions of the HIV-1 proteome into one chimaeric protein. This gene has been inserted into 2 leading non-replicating vaccine vectors: an attenuated chimpanzee adenovirus serotype 63 (ChAdV63) and a modified vaccinia virus Ankara (MVA) to construct the ChAdV63.HIVconsv and MVA.HIVconsv HIV-1 candidate vaccines. The present study is named ChAd-MVA.HIVconsv-BCN01 and it is a phase I, multicenter primary/booster therapeutic vaccination study to evaluate the safety and immunogenicity of ChAdV63.HIVcons and MVA.HIVconsv HIV-1 vaccines, delivered intramuscularly according to a 0-8 weeks or a 0-24 weeks schedule to recently HIV-1 infected individuals with early viral suppression 6 months after initiation of Tenofovir/Emtricitabine plus Raltegravir.

DETAILED DESCRIPTION:
It is a Phase I, multicenter primary/booster therapeutic vaccination study to evaluate the safety and immunogenicity of ChAdV63.HIVcons and MVA.HIVconsv HIV-1 vaccines, delivered intramuscularly according to a 0-8 weeks or a 0-24 weeks schedule to recently HIV-1 infected individuals with early viral suppression 6 months after initiation of Tenofovir/Emtricitabine plus Raltegravir.

24 patients who meet all eligibility criteria will be enrolled, first 10 individuals will be assigned in the 0-24 week prime/boost regimen (ARM A). The next 10 volunteers will be assigned in the 0-8 week prime/boost regimen (ARM B).Four additional volunteers will be included as 'back-up' and assigned 2 in ARM A and 2 in ARM B to cover a possible 10% of patients who drop-off during the follow-up. Purpose of staging of 2 study arms is just to shorten overall study duration (from screening of first volunteer to 6 months after last immunisation of last volunteer).

Lastly, 24 patients who also meet all eligibility criteria will be enrolled as controls, will also initiate promptly antiretroviral treatment with Tenofovir/Emtricitabine plus Raltegravir but will not receive the investigational vaccines. Control patients will consecutively be assigned to the 0-24w control arm (ARM C 'long control') or 0-8w control arm (ARM D 'short control') until 12 patients per arm are reached. The purpose of the control arms is to have a study population to compare the viral reservoir decay kinetics in the absence of vaccination.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, aged 18-60 years
2. Confirmed HIV-1 seropositive documented in the past 6 months (by acute antiretroviral syndrome, p24 antigenemia and/or ELISA seroconversion)
3. Willing and able to give written informed consent for participation in the study
4. Willing and able to adhere to an effective HAART regimen for the duration of the study
5. Cluster of differentiation 4 (CD4)+ T cell count > 350 cells/ml at screening and at the preceding clinic visit
6. No new AIDS-defining diagnosis or progression of HIV-related disease.
7. Haematological and biochemical laboratory parameters as follows: Haemoglobin > 10g/dl, Platelets > 100.000/dl, alanine aminotransferase (ALT) ≤ 2.5 x ULN, Creatinine ≤ 1.3 x upper limit of normal (ULN)
8. Serology: negative for hepatitis B surface antigen OR HbsAg positive with Hepatitis B Virus (HBV)-DNA < 1000 copies/ml; negative for hepatitis C antibodies OR confirmed clearance of Hepatitis C Virus (HCV) infection (spontaneous or following treatment); negative syphilis serology or documented adequate treatment of syphilis if positive enzimeimmunoassay (EIA) Immonoglobulin G (IgG) or Treponema pallidum hemagglutination assay (TPHA)
9. Available for follow up for duration of study (screening + 72 weeks) and willing to comply with the protocol requirements
10. Women of child-bearing age must not be pregnant, not be planning a pregnancy or breast-feeding. Sexually active women must be willing to use an approved method of contraception from screening until 4 months after the second immunisation. Sexually active men in heterosexual relationships must be willing to use an approved method of contraception with their partners from screening until 4 months after the second immunisation.

Exclusion Criteria:

1. Confirmed HIV-2 seropositive
2. Positive pregnancy test
3. Presence of Nucleos(t)ide Reverse Transcriptase Inhibitors (NRTI) mutation in the screening genotype
4. Participation in another clinical trial within 12 weeks of study entry
5. History of autoimmune disease other than HIV-related auto-immune disease.
6. History or clinical manifestations of any physical or psychiatric disorder which could impair the subject's ability to complete the study
7. History of anaphylaxis or severe adverse reaction to vaccines
8. Previous immunisation with any experimental immunogens
9. Receipt of blood products within 6 months of study entry
10. Treatment for cancer or lymphoproliferative disease within 1 year of study entry
11. Receipt of vaccines other than Hepatitis B vaccine within 2 weeks of study entry or planned receipt within 2 weeks of vaccination
12. Any other prior therapy which, in the opinion of the investigators, would make the individual unsuitable for the study or influence the results of the study
13. Current or recent use (within last 3 months) of interferon or systemic corticosteroids or other immunosuppressive agents

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2012-10; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Grade 3 or 4 local reaction | Up to 24 weeks
  The proportion of volunteers who develop a grade 3 or 4 local reaction
Grade 3 or 4 systemic reaction | Up to 24 weeks
  The proportion of volunteers who develop a grade 3 or 4 systemic reaction
Serious adverse event, including laboratory abnormalities. | Up to 24 weeks
  The proportion of volunteers who develop a serious adverse event, including laboratory abnormalities.

SECONDARY OUTCOMES:
HIV-specific CD8+ T cell responses | Change from baseline (pre-HAART) and w24, to +1week, +4weeks, +12weeks and +24weeks post vaccination.
  Magnitude and phenotype of HIV-1-specific CD8+ T cell populations , in selected volunteers with appropriate human leukocyte antigen (HLA) class I alleles will be assessed according to first immunogenicity results.
Magnitude and phenotype of HIV-1-specific CD8+ T cell populations | Change from baseline (pre-HAART) and w24, to +1week, +4weeks, +12weeks and +24weeks post vaccination.
  Magnitude and phenotype of HIV-1-specific CD8+ T cell populations , in selected volunteers with appropriate HLA class I alleles will be assessed according to first immunogenicity results.
Lymphocyte activation marker HLADR+CD38+ | Change from baseline (pre-HAART) and w24, to +1week, +4weeks, +12weeks and +24weeks post vaccination.
  Lymphocyte activation marker HLA-DR+CD38+ will be assessed at selected timepoints according to first immunogenicity results
Integrated and unintegrated viral HIV-1 DNA in PBMCs. | Change from baseline (pre-HAART) and w24, to +1week, +4weeks, +12weeks and +24weeks post vaccination.
  Quantification of integrated and unintegrated viral HIV-1 DNA in peripheral blood mononucleated cells (PBMC)s will be determined at selected timepoints according to first immunogenicity results
Viral suppressive capacity of CD8+ T cells in vitro | Change from baseline (pre-HAART) and w24, to +1week, +4weeks, +12weeks and +24weeks post vaccination.
  Viral suppressive capacity of CD8+ T cells in vitro using a flow cytometric assay at selected timepoints according to first immunogenicity results

CONTACTS AND LOCATIONS:
Overall Officials: Christian Brander, PhD, Study Chair — Institut de Recerca de la Sida IrsiCaixa-HIVACAT; Beatriz Mothe, MD,PhD, Principal Investigator — Institut de Recerca de la Sida IrsiCaixa-HIVACAT; Josep Maria Miró, MD,PhD, Principal Investigator — Hospital Clínic i Provincial de Barcelona, HIVACAT
Locations (2):
- Spain (2):
  - Germans Trias i Pujol Hospital, Badalona, Barcelona
  - Clinic de Barcelona Hospital, Barcelona

REFERENCES:
- [Derived] Mothe B, Manzardo C, Sanchez-Bernabeu A, Coll P, Moron-Lopez S, Puertas MC, Rosas-Umbert M, Cobarsi P, Escrig R, Perez-Alvarez N, Ruiz I, Rovira C, Meulbroek M, Crook A, Borthwick N, Wee EG, Yang H, Miro JM, Dorrell L, Clotet B, Martinez-Picado J, Brander C, Hanke T. Therapeutic Vaccination Refocuses T-cell Responses Towards Conserved Regions of HIV-1 in Early Treated Individuals (BCN 01 study). EClinicalMedicine. 2019 Jun 5;11:65-80. doi: 10.1016/j.eclinm.2019.05.009. eCollection 2019 May-Jun. PMID 31312806